CLINICAL TRIAL: NCT01762813
Title: Prospective, Population-based Cohort Collection of Blood Samples and Tumor Tissue From Patients Operated on for Primary or Metastatic Colorectal Cancer
Brief Title: Assessment of Clinically Related Outcomes and Biomarker Analysis for Translational Integration in Colorectal Cancer
Acronym: ACROBATICC
Status: Recruiting | Type: Observational
Sponsor: Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Other Study IDs: 29034/2012
Record Dates: First submitted 2013-01-03; First posted 2013-01-08 (Estimated); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Colorectal Cancer
Keywords: Colon cancer; rectal cancer; liver metastasis; survival; biomarker; molecular profile
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, whole blood, plasma, cancer tissue, normal tissue.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- open and laparoscopic surgery: Patients with primary and or metastatic colorectal cancer (CRC) eligible for curative surgery will be included. Subcohorts may be based on either colon cancer, rectal cancer, metastatic cancer, surgery (laparoscopy or open), node negative and node positive disease, and molecular profiling.
  Interventions: Procedure: open and laparoscopic surgery

INTERVENTIONS:
Procedure: open and laparoscopic surgery — Curative surgery for either primary (colorectal cancer, crc) or metastatic CRC (liver surgery)
  Other Names: Liver surgery

SUMMARY:
* A prospective, observational study on clinical outcomes of surgical management of primary and metastatic colorectal cancer
* Prospective collection of tissues to explore potential biomarkers in blood and/or primary or secondary cancers and/or normal colon

DETAILED DESCRIPTION:
Prospective project in collecting and assessing clinical outcomes data related to molecular profiling of tumors based on cancer primary or metastatic tissue or tissue from peripheral blood samples. As a future part of the project will be collected patient reported outcomes (PROs) for assessing clinical outcomes in relation to clinical pathways, patient reported results, as well as tumor profiling by molecular methods.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of colorectal cancer, primary or metastatic (liver), with a treatment intention of planned curative surgery
* Informed consent to participate
* Age ≥18

Exclusion Criteria:

* failure to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with colorectal cancer (primary and/or secondary) undergoing surgery for curative intent
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2013-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Cancer-specific survival | 5-years
  Time from surgery to death of cancer

SECONDARY OUTCOMES:
Recurrence-free survival | 3 and 5 years
  Time from surgery to recurrence of cancer

CONTACTS AND LOCATIONS:
Overall Officials: Kjetil Søreide, MD, PhD, FRCS, FACS, Principal Investigator — Helse Stavanger HF
Locations (1):
- Stavanger University Hospital, Stavanger, Norway

IPD SHARING:
Plan to Share IPD: Undecided
Raw data may be provided given appropriate consent and approval for anonymous database sharing

REFERENCES:
- [Background] Soreide K, Watson MM, Lea D, Nordgard O, Soreide JA, Hagland HR; ACROBATICC collaborators. Assessment of clinically related outcomes and biomarker analysis for translational integration in colorectal cancer (ACROBATICC): study protocol for a population-based, consecutive cohort of surgically treated colorectal cancers and resected colorectal liver metastasis. J Transl Med. 2016 Jun 29;14(1):192. doi: 10.1186/s12967-016-0951-4. PMID 27357108
- [Result] Hagland HR, Lea D, Watson MM, Soreide K. Correlation of Blood T-Cells to Intratumoural Density and Location of CD3+ and CD8+ T-Cells in Colorectal Cancer. Anticancer Res. 2017 Feb;37(2):675-683. doi: 10.21873/anticanres.11363. PMID 28179316
- [Result] Watson MM, Lea D, Hagland HR, Soreide K. Elevated Microsatellite Alterations at Selected Tetranucleotides (EMAST) Is Not Attributed to MSH3 Loss in Stage I-III Colon cancer: An Automated, Digitalized Assessment by Immunohistochemistry of Whole Slides and Hot Spots. Transl Oncol. 2019 Dec;12(12):1583-1588. doi: 10.1016/j.tranon.2019.08.009. Epub 2019 Oct 31. PMID 31677491
- [Result] Watson MM, Kanani A, Lea D, Khajavi RB, Soreide JA, Korner H, Hagland HR, Soreide K. Elevated Microsatellite Alterations at Selected Tetranucleotides (EMAST) in Colorectal Cancer is Associated with an Elderly, Frail Phenotype and Improved Recurrence-Free Survival. Ann Surg Oncol. 2020 Apr;27(4):1058-1067. doi: 10.1245/s10434-019-08048-6. Epub 2019 Nov 4. PMID 31686344
- [Result] Lea D, Zaharia C, Soreide K. Programmed death ligand-1 (PD-L1) clone 22C3 expression in resected colorectal cancer as companion diagnostics for immune checkpoint inhibitor therapy: A comparison study and inter-rater agreement evaluation across proposed cut-offs and predictive (TPS, CPS and IC) scores. Cancer Treat Res Commun. 2024;38:100788. doi: 10.1016/j.ctarc.2023.100788. Epub 2023 Dec 22. PMID 38150845
- [Result] Watson MM, Lea D, Gudlaugsson E, Skaland I, Hagland HR, Soreide K. Prevalence of PD-L1 expression is associated with EMAST, density of peritumoral T-cells and recurrence-free survival in operable non-metastatic colorectal cancer. Cancer Immunol Immunother. 2020 Aug;69(8):1627-1637. doi: 10.1007/s00262-020-02573-0. Epub 2020 Apr 20. PMID 32314040
- See also: ACROBATICC protocol paper — http://www.ncbi.nlm.nih.gov/pubmed/27357108
- Available data/document: Study Protocol — http://translational-medicine.biomedcentral.com/articles/10.1186/s12967-016-0951-4